CLINICAL TRIAL: NCT04677127
Title: The Effect of Health Belief Model and Health Literacy Level Based Education and Counseling on Glycemic Control in Type 2 Diabetes Patients
Brief Title: Effect of HBM Based Education on Glycemic Control of Type 2 Diabates Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, İmatullah Akyar, Associate professor, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 16969557-1072
Record Dates: First submitted 2020-12-14; First posted 2020-12-21 (Actual); Last update posted 2020-12-21 (Actual); Status verified 2020-12

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Health Belief Model; Counseling

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): The intervention group was given training based on the health belief model with groups of 10-12-13 people every week for 6 weeks in the Family Health Center, followed by telephone counseling in the following 6 weeks and follow-up for 12 weeks.
  Interventions: Behavioral: Health Belief Model and Health Literacy Level based Education and Counseling
- Control (No Intervention): Patients in the control group were assessed at the first interview and the last interview, received routine health care, and no intervention was performed during the research.

INTERVENTIONS:
Behavioral: Health Belief Model and Health Literacy Level based Education and Counseling — Patients given education and counseling constructed with health belief model (perceived susceptibility, perceived severity, perceived benefits, perceived barriers, cue to action, self-efficacy). The constructed education given through groups dichotomised by health literacy levels (low/high). Groups of 11-13, had weekly educations for 6 weeks, 6 weeks of counselling and 12 week of follow-up.
  Arms: Intervention

SUMMARY:
This pre-post-test randomized controlled (parallel group) experimental design study aimed to determine the effect of education based on health belief model and health literacy level of patients with type 2 diabetes on disease management. Study was carried out in Isparta Davraz Family Health Centre between June 17, 2019 and March 02, 2020. Sample consisted of 120 patients with type 2 diabetes, selected by simple randomization method, including 60 patients for the intervention group and 60 patients for the control group.

Patients in intervention and control were also sub-grouped according to their health literacy level. The intervention group was given training based on the health belief model with groups of 10-12-13 people every week for 6 weeks in the Family Health Center, followed by telephone counseling in the following 6 weeks and follow-up for 12 weeks. Patients in the control group were assessed at the first interview and the last interview, received routine health care, and no intervention was performed during the research. "Patient Data Form", "Health Literacy Scale Among Diabetes Patients", "Health Belief Model Scale in Diabetes Patients" and "Type 2 Diabetes Self-Efficacy Scale" used for data collection. Data were collected both on the first day of the study and in the 24th week.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of type 2 Diabates Mellitus at least for a year
* Literate

Exclusion Criteria:

* Problems with vision and hearing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2019-06-17 (Actual); Primary Completion 2020-03-02 (Actual); Study Completion 2020-03-02 (Actual)

PRIMARY OUTCOMES:
Glycemic Control Change | pre-test (week 1), post-test (week 24)
  HbA1C-Change from Baseline HbA1C at 6 months

SECONDARY OUTCOMES:
Health Belief Model Questionnaire | pre-test (week 1), post-test (week 24)
  Change in perceived severity, perceived susceptibility, perceived benefits, perceived barriers scores
Self-Efficacy Questionnaire | pre-test (week 1), post-test (week 24)
  Change from Baseline self-efficacy level scores at 6 months

CONTACTS AND LOCATIONS:
Overall Officials: İmatullah Akyar, Principal Investigator — Hacettepe University
Locations (1):
- Hacettepe University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Agrali H, Akyar I. The effect of health literacy-based, health belief-constructed education on glycated hemoglobin (HbA1c) in people with type 2 diabetes: A randomized controlled study. Prim Care Diabetes. 2022 Feb;16(1):173-178. doi: 10.1016/j.pcd.2021.12.010. Epub 2021 Dec 31. PMID 34980562